CLINICAL TRIAL: NCT02792634
Title: Pathogenesis of Non-alcoholic Steatohepatitis and Liver Regeneration After Bariatric Surgery / Untersuchung Der Pathogenese Der Nicht-alkoholischen Steatohepatitis Und Der Leberregeneration Nach Bariatrischer Chirurgie
Brief Title: Pathogenesis of Non-alcoholic Steatohepatitis and Liver Regeneration After Bariatric Surgery
Acronym: NALKOSTEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-164
Record Dates: First submitted 2016-03-22; First posted 2016-06-07 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-05

CONDITIONS: Bariatric Surgery Candidate; Nonalcoholic Steatohepatitis; Obesity
Keywords: Bariatric surgery; Nonalcoholic Steatohepatitis; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sleeve-Gastrectomy, Roux en Y gastric bypass

SUMMARY:
Obesity and obesity related health problems are globally recognized as one of the major threats to public health. Bariatric surgery is the most effective and durable therapy option for obesity and the improvement of obesity related co-morbidities. "Non alcoholic steatohepatitis" (NASH) is an important comorbidity of obesity and improves after surgical intervention. In this study investigators try to enlighten the weight independent mechanism for the effects of bariatric surgery. Patients who are assigned to a bariatric procedure will be observed for at least 24 month. A liver and adipose tissue samples are gained during the operation. Liver function and morphology are observed before and after operation with LiMAx, FibroScan and ultrasound. Systemic inflammation is measured in blood samples before and after surgical intervention. In order to check the microbiome stool samples are collected throughout the entire observation period.

DETAILED DESCRIPTION:
Every patient who is scheduled for bariatric surgery in the university hospital Aachen will be evaluated for this study. After informed consent baseline measurements are performed preoperative. Baseline measurements involve blood and stool samples, LiMAx, FibroScan and ultrasound. During the operation a liver, a subcutaneous and visceral fat sample are taken to analyse liver histology and inflammation as well as fatty tissue signaling. After the operation patients are observed 24 month. Further blood samples are taken on the first postoperative day, 2 and 4 weeks, 3, 6, 12, 18 and 24 month after the operation. Stool samples are taken 2 and 4 weeks, 3, 6, 12, 18 and 24 month after the intervention. The LiMAx test, a test analysing the liver function, is performed 4 weeks, 6, 12 and 24 month after the operation. The morphologic liver structure is evaluated by FibroScan and ultrasound 4 weeks, 6, 12 and 24 month postoperative.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* scheduled for bariatric surgery
* informed consent

Exclusion Criteria:

* pregnancy
* substance abuse
* liver disease other than NASH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BMI > 35 kg/m2 Age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Weight in kg | 24 month

SECONDARY OUTCOMES:
NAFLD (Non-alcoholic fatty liver disease) Activity Score (NAS) | within 7 days after the operation
  The NAS will be assessed by a trained pathologist in a liver sample which is taken during the operation. The NAS usually will be assessed within 7 days after the Operation. The NAS is the basis for further clinical and laboratory tests and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany